CLINICAL TRIAL: NCT06586866
Title: A Multicenter, Single-Arm, Phase 2 Study to Evaluate the Safety, Efficacy and Pharmacokinetics of JK-1201I in Triple Negative Breast Cancer Patients with Brain Metastases
Brief Title: JK-1201I in Triple Negative Breast Cancer Patients with Brain Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: JenKem Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JK-1201I-203
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Triple Negative Breast Cancer (TNBC); Brain Metastasases
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JK-1201I (Experimental): Participants will receive JK-1201I as an intravenous (IV) infusion at dose of 125mg/m2 on Day 1 of each 14-day cycle until a treatment discontinuation criterion is met as specified in the protocol.
  Interventions: Drug: JK-1201I

INTERVENTIONS:
Drug: JK-1201I — JK-1201I will be administered as an IV infusion at dose of 125mg/m2 on Day 1 of each 14-day cycle.

SUMMARY:
This study was designed to evaluate the safety, efficacy and pharmacokinetics of JK-1201I in triple negative breast cancer patients with brain metastases.

DETAILED DESCRIPTION:
This is a multicenter, single-arm, phase 2 study to evaluate the safety, efficacy and pharmacokinetics of JK-1201I in triple negative breast cancer patients with brain metastases.

Patients will receive JK-1201I until disease progression. The primary objective of this study is to assess whether treatment with JK-1201I prolongs progression-free Survival (PFS) according to RECIST 1.1 and RANO-BM in triple negative breast cancer patients with brain metastases.

The secondary objectives of the study are to further evaluate the efficacy, safety and pharmacokinetics of JK-1201I.

ELIGIBILITY:
Inclusion

Participants must meet all the following criteria to be eligible for randomization into the study:

1. Sign and date the informed consent form prior to the start of any study-specific qualification procedures.
2. Female aged ≥18 years.
3. Has ECOG PS of ≤1.
4. Life expectancy ≥ 3months.
5. Histological or cytological confirmation of triple-negative breast cancer (TNBC).
6. At least one prior chemotherapy regimen with anthracyclines and taxanes for advanced disease.
7. Has at least 1 measurable brain metastatic lesion according to RANO-BM.
8. Adequate biological function.
9. Men or women should be using adequate contraceptive measures during the study and for 6 months following the last dose of investigational product.

Exclusion

Participants who meet any of the following criteria will be disqualified from entering the study:

1. Patients who have received prior anti-cancer treatment within 4 weeks.
2. . Patients must not have previously received JK-1201I or any other form of irinotecan, SN38.
3. Hypersensitivity to any ingredient of JK-1201I and Topotecan.
4. Current use or any use in the last two weeks of strong CYP3A-enzyme inducers / in the last two weeks of strong CYP3A-enzyme inhibitors and / or strong UGT1A inhibitors.
5. Unresolved toxicity from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 1 with exceptions defined in the protocol.
6. History of other malignancies within last 5 years.
7. History of immunodeficiency disease, or positive human immunodeficiency virus antibody.
8. Severe infections within 4 weeks before the first use of the study drug.
9. Active hepatitis B virus infection, or active hepatitis C virus infection.
10. Patients who received surgery within last 4 weeks before the initiation of study treatment.
11. Patients with brain stem, meningeal or spinal cord metastasis.
12. Severe symptoms by tumor aggressive important organ.
13. Uncontrolled hydrothorax and ascites.
14. Uncontrolled concomitant systemic disorder as defined in the protocol.
15. Serious cardiac condition or uncontrolled high blood pressure.
16. History of mental illness, drug abuse, alcoholism.
17. Pregnant or breast-feeding.
18. Other conditions that the investigator considers unsuitable to participate in this clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 25 (Estimated)
Dates: Start 2024-09-26 (Estimated); Primary Completion 2026-05-26 (Estimated); Study Completion 2026-10-26 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) according to RECIST 1.1 and RANO-BM | Up to approximately 12 months.
  Progression-free Survival (PFS) is defined as the time interval from the randomization to disease progression or death due to any cause.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) according to RECIST 1.1 | Up to approximately 12 months.
  Progression-free Survival (PFS) is defined as the time interval from the randomization to disease progression or death due to any cause.
Progression-free Survival (PFS) according to RANO-BM | Up to approximately 12 months.
  Progression-free Survival (PFS) is defined as the time interval from the randomization to disease progression or death due to any cause.
Objective Response Rate (ORR) according to RECIST 1.1 | Up to approximately 6 months.
  Confirmed ORR is defined as the proportion of participants who have achieved a best overall response of confirmed complete response (CR), confirmed partial response (PR) according to RECIST 1.1.
Objective Response Rate (ORR) according to RANO-BM | Up to approximately 6 months.
  Confirmed ORR is defined as the proportion of participants who have achieved a best overall response of confirmed complete response (CR), confirmed partial response (PR) according to RANO-BM.
Overall survival (OS) | Up to approximately 24 months.
  Overall survival (OS) is defined as the time interval from randomization to death due to any cause.
Incidence and Grade of Participants with Adverse Events or Serious Adverse Events | Up to approximately 24 months.
  Adverse Events (AEs) or Serious Adverse Events (SAEs) are assessed based on NCI CTCAE v5.0.
Pharmacokinetic Parameter Area Under the Plasma Concentration-Time Curve for JK-1201I, Irinotecan, SN38 and SN38G | Up to 6 months.
  Area under the plasma concentration-time curve up to the last quantifiable time point (AUClast) and area under the plasma concentration-time curve dosing interval (AUCtau) will be assessed using Non-linear mixed effect modeling.
Pharmacokinetic Parameter Maximum Concentration for JK-1201I, Irinotecan, SN38 and SN38G | Up to 6 months.
  Maximum concentration (Cmax) will be assessed using Non-linear mixed effect modeling.